## Graftless Closed Sinus Tenting Using Dental Implants After Densah Burs Osteotomy Versus Conventional Osteotomy in Localized Sinus Pneumatization: a Randomized Clinical Trial

Thesis Protocol Submitted for Partial Fulfillment of the Requirements for Master's Degree In Oral & Maxillofacial Surgery Faculty of Oral & Dental Medicine - Cairo University

By

Basma Mohammed Shaheen
B.D.S Oral & Dental Medicine, MIU Uni. 2016, Egypt

(26th October, 2021)

**Code: OMFS 3-3-5** 

3000

## Medical Biostatistics Unit review report for sample size calculation

Researcher's Full name: Basma Mohammed Shaheen

Email address: basma.shaheen@icloud.com

Degree: Master Postgraduate Student

Department: Oral and Maxillofacial Surgery

Main Supervisor details (if applicable)

Full name: Prof. Dr. Sameh Mekhemer

Email address

Research title: Graftless Closed Sinus Tenting Using Dental Implants After Densah Bur Osteotomy Versus Conventional Osteotome in Localized Sinus Pneumatization. A Randomized Clinical Trial.

Research question: Will the use of densah bur lead to better bone gain around implant than conventional dosed sinus lift in isolated pneumatized sinus?

## Items used in the calculated sample size

- The outcome used (State 1ry or 2ry):bone gain
- Values used for outcome (e.g. mean difference, percentage, proportion..... etc.)
- Entry 1: (mean difference between 2 groups, mean and standard deviation of group 1, proportion 1 or estimated prevalence) = 9.93±0.57.
  - Entry 2: (standard deviation of control group, mean and standard deviation of group 2, proportion 2 or clinically important difference)= 10.71±0.43.
- Alpha level of significance:0.05
- Effect size used in calculation:1.544
- Power of the study:80%
- Statistical test used:Independent-t-test
- The calculated sample size: 8 per group, total=16 patients
- Increased number for anticipated missing data: 15% to compensate for drop outs, 10 per group, total=20 patients.

## Decision of MBU:

| • | Accepted* |
|---|----------------------|
| • | Needs modifications |
| | What to be modified: |
| | A meeting is needed |

Date of meeting: / /

Time of meeting:

Place of meeting:

N.B. If you couldn't attend the meeting, show up to apologize or contact your reviewer by email to set up another convenient time.

MBU member

Ass Prof Nouran AbdelNabi

MBU Director

Prof Dr Noha Ghallab

\* Date of submission: 13 / 9 / 2021

Date of approval: 22 / 9 /2021

Vice Dean for Postgraduate affairs and research